CLINICAL TRIAL: NCT01906723
Title: Evaluation of the Effectiveness of a Novel Gait Trainer in Increasing the Functionality of Motor Impaired Patients: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Purpose: Supportive Care
Other Study IDs: UpnFree-HMO-CTIL
Record Dates: First submitted 2013-07-21; First posted 2013-07-24 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2013-07

CONDITIONS: To Evaluate Effectiveness of the Gait Trainer in Increasing the Functionality and Spatiotemporal Parameters of Gait of 4 Patients.
MeSH Terms: interventions — Walkers

INTERVENTIONS:
Device: Walker — The Up n' Free (Easy Walking) is a gait trainer equipped with a dynamic partial weight-bearing. The trainer is designed to provide the user with independence, safety, and endurance. It allows for easy transfer from sitting to standing position and stabilizes the pelvis, allowing for free movement of the hands.
  Other Names: Up n' Free trainer

SUMMARY:
Unstrained ambulation is the main goal of gait rehabilitation for preventing fatigue and increasing functionality in patients with gait deficiencies. The Up n' Free (Easy Walking) is a gait trainer equipped with a dynamic partial weight-bearing. The trainer is designed to provide the user with independence, safety, and endurance. It allows for easy transfer from sitting to standing position and stabilizes the pelvis, allowing for free movement of the hands. The effectiveness of the Up n' Free trainer in increasing the patient's functionality at the hospital or at home has not been quantified. We therefore aim to evaluate effectiveness of the gait trainer in increasing the functionality and spatiotemporal parameters of gait of 4 patients.

DETAILED DESCRIPTION:
Four ambulatory adults with postpolio syndrome, multiple sclerosis, cerebral palsy and spinal cord injury will be recruited for the study (one of each pathology).

Inclusion criteria:

* Ambulatory patients ages of 18 and above
* Cognitive and cooperative ability to follow simple instructions
* Independently capable to understand an informed consent form
* Weight below 100kg

Exclusion criteria:

• Cognitive disorders preventing the subject from understanding the trial protocol or following the researcher's instructions

2.2 Trial Protocol The subjects will be recruited from the rehabilitation department at the Hadassah medical center. Each subject will understand and agree to an informed consent form pretrial. The subjects' age, weight, and BMI will be documented. They will then receive a 10- minutes instruction on using the Up n' Free gait trainer and will be provided with the trainer for the 1-week duration of the trial. Spatiotemporal parameters and gait symmetry will be recorded in the Hadassah gait laboratory, while the patient ambulates with his or her own walking aid. Physical Activity (PA) will be assessed using triaxial accelerometer-based activity monitors (ActiGraph GT3X, Pensacola, Florida, USA), using a preset sampling epoch of 1s. The participants will be instructed to wear the activity monitors on their right hip for 7 consecutive days and only remove it during night time sleep or water activities. At the end of 7 days the subjects will return the Up n' Free gait trainer and fill out a satisfactory questionnaire. Spatiotemporal parameters and gait symmetry will be recorded again in the Hadassah gait laboratory, while the patient ambulates with the Up n' Free.

2.3 Data Analysis Estimates of the PA will be weighed by 5/7th of the weekly activity for the weekdays (Sunday-Thursday) and 2/7th for weekend days (Friday and Saturday) as within-week variation is expected. Total PA (1,000 counts × day-1), wear time PA (count × min-1), sedentary time (hours × day-1; between 0-99 counts/min), low-light PA (min×day-1; between 100-759 counts/min), High-light PA (min × day-1; 760-2019 counts/min), moderate-vigorous PA (min × day-1; ≥2020 counts/min).

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients ages of 18 and above
* Cognitive and cooperative ability to follow simple instructions
* Independently capable to understand an informed consent form
* Weight below 100kg

Exclusion Criteria:

* Cognitive disorders preventing the subject from understanding the trial protocol or following the researcher's instructions

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Physical activity | 1 week
  Activity monitor data (via accelerometers)

SECONDARY OUTCOMES:
Spatio-temporal parameters | baseline, 1 week following baseline
  step length, gait velocity, stance duration

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel